CLINICAL TRIAL: NCT05766904
Title: Efficacy of a Meningococcal B Vaccine Against Neisseria Gonorrhoeae Infections Among Men Who Have Sex With Men: a Randomised-controlled Clinical Trial
Brief Title: Efficacy Trial on Meningococcal B Vaccine for Preventing Gonorrhea Infections
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Tsz Ho Kwan, Research Assistant Professor, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 21200912
Record Dates: First submitted 2023-03-01; First posted 2023-03-13 (Actual); Last update posted 2025-04-04 (Actual); Status verified 2025-04

CONDITIONS: Gonorrhea; Sexually Transmitted Infection
MeSH Terms: conditions — Gonorrhea; Sexually Transmitted Diseases | interventions — 4CMenB vaccine

STUDY DESIGN:
Intervention Model Description: Participants in the vaccination group would receive two doses of 4CMenB vaccine 1 month apart (at Month 0 and Month 1) while subjects in the control group would receive two doses of normal saline of a similar volume.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Block randomisation would be used to generate the list of treatment groups with a block size of 4 in a centralised computer by a staff in the Research Centre unrelated to data analysis. Group assignment would be concealed and performed by another staff unrelated to data analysis who will pick the group number from the random allocation sequence in sequential order. The subjects and investigators would therefore be blinded.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention (Experimental): Intramuscular injection of 2 doses of 0.5mL 4CMenB vaccine 1 month apart
  Interventions: Biological: 4CMenB vaccine
- Control (Placebo Comparator): Intramuscular injection of 2 doses of 0.5mL placebo 1 month apart
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: 4CMenB vaccine — Four-component MenB vaccine
  Other Names: Bexsero
  Arms: Intervention
Other: Placebo — 0.9% Sodium Chloride Inj. B.P.
  Arms: Control

SUMMARY:
Objectives: Efficacy of a meningococcal vaccine against Neisseria gonorrhoea (NG) infection among men who have sex with men (MSM).

Design: Parallel randomised double-blind placebo-controlled trial.

Setting: A teaching hospital in Hong Kong.

Participants: 150 adult MSM at risk of gonorrhoea infection (condomless sex with more than one man within the last six months, history of sexually transmitted infection [STI] diagnosis, inclination to have condomless sex, and other PrEP-eligible criteria) would be recruited into the trial, with half allocated to intervention and control group each.

Intervention: Intervention and control group would receive, one month apart, two doses of meningococcal vaccine and normal saline, respectively.

Main outcome measures: Safety and efficacy of vaccine against gonorrhoea (time to first gonorrhoea infection and incidence), and behavioural change after vaccination.

Expected results: NG incidences in two groups would be compared. Efficacy of vaccine against gonorrhoea would be determined after controlling confounding variables. Characteristics of participants with incident NG would be distinguished from those without incident infections. Change of frequency of sexual activities and networking would be noted.

Implications: Strategies on STI screening and vaccination could be informed. Reduced STI burden post-vaccination could be measured with surveillance system.

ELIGIBILITY:
Inclusion Criteria:

* Male adult who has had sex with another male in the past six months
* Ages 18 years or above
* Normally resides in Hong Kong
* Able to communicate in written and spoken Chinese or English
* At risk of gonorrhoea infection (had condomless sex with more than one man within the last six months, history of STI diagnosis, inclination to have condomless sex, and other PrEP-eligible criteria)
* Negative NG test result at the time of recruitment
* No history of previous vaccination with MenB vaccines
* Able and willing to attend all study visits

Exclusion Criteria:

* Contraindications to receive MenB vaccine
* Unable to give informed consent

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 150 (Estimated)
Dates: Start 2023-05-04 (Actual); Primary Completion 2025-09 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Comparison between incidence of NG between two groups | Month 2 to Month 24
  Difference in NG incidences in the two groups

SECONDARY OUTCOMES:
Changes in risk behaviours and networking pattern after vaccination | Month 2 to Month 24
  Frequency of sex networking, number of sex partners, and use of condoms
Safety profile of the vaccine | Month 2 to Month 24
  Prevalence of adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Tsz Ho Kwan, PhD, Principal Investigator — Jockey Club School of Public Health and Primary Care
Locations (1):
- Stanley Ho Centre for Emerging Infectious Diseases, Shatin, Hong Kong